CLINICAL TRIAL: NCT06430268
Title: Efficacy of Non-surgical and Surgical Surface Decontamination Methods on Peri-implantitis-affected Implants: A Randomized Clinical Trial
Brief Title: Efficacy of Non-surgical and Surgical Surface Decontamination Methods on Peri-implantitis-affected Implants
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Andrea Ravida (Other)
Collaborators: Association for Dental Infection Control (Unknown)
Responsible Party: Sponsor-Investigator, Andrea Ravida, Assistant Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY23100029
Record Dates: First submitted 2024-05-21; First posted 2024-05-28 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Peri-Implantitis; Dental Implant Failed
Keywords: Peri-implantitis; Decontamination; Implant Surface
MeSH Terms: conditions — Peri-Implantitis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (5):
- Non-surgical decontamination with titanium curettes followed by explantation (Experimental): Titanium curettes (Hu-Friedy, Chicago, Illinois, USA) will be used for supra and submucosal around the implants without any flap elevation.
  Interventions: Procedure: implant decontamination with titanium curette
- Non-surgical decontamination with erythritol powder prior to implant removal (Experimental): Without any flap elevation, the supramucosal implant surfaces will be cleaned with the Airflow handpiece, while for the submucosal areas, a Perioflow handpiece and nozzle for submucosal instrumentation will be used. The nozzle will be changed after cleaning each implant.
  Interventions: Device: implant decontamination with Air-Flow device
- Surgical decontamination with titanium curettes prior to implant removal (Experimental): Intra-sulcular and, if necessary, vertical releasing incisions will be performed. Full-thickness flaps will be elevated in the buccal and lingual aspects and the granulation tissue will be removed. Titanium curettes (Hu-Friedy, Chicago, Illinois, USA) will be used for supra and submucosal around the implants
  Interventions: Procedure: implant decontamination with titanium curette
- Surgical decontamination with erythritol powder prior to implant removal (Experimental): Intra-sulcular and, if necessary, vertical releasing incisions will be performed. Full-thickness flaps will be elevated in the buccal and lingual aspects and the granulation tissue will be removed.The Airflow handpiece will be moved in a horizontal direction along implant threads from an apical to a coronal position. The angulation of the handpiece and working distance will not be standardized as they may vary according to the area being cleaned.
  Interventions: Device: implant decontamination with Air-Flow device
- No decontamination prior to implant removal (No Intervention): No decontamination will be performed on implants in this group.

INTERVENTIONS:
Procedure: implant decontamination with titanium curette — Titanium curettes (Hu-Friedy, Chicago, Illinois, USA) will be used for supra and submucosal around the implant, with and without flap elevation.
  Arms: Non-surgical decontamination with titanium curettes followed by explantation; Surgical decontamination with titanium curettes prior to implant removal
Device: implant decontamination with Air-Flow device — Air-polishing (Airflow Prophylaxis Master, EMS, Nyon, Switzerland) will be carried out with AIR-FLOW powder PLUS (EMS) containing erythritol (sugar alcohol, 14 μm), amorphous silica and 0.3% chlorhexidine to decontaminate implants with and without flap elevation. The device will be adjusted to a power setting of 5 bar static pressure and a maximum level of irrigation with water.
  Arms: Non-surgical decontamination with erythritol powder prior to implant removal; Surgical decontamination with erythritol powder prior to implant removal

SUMMARY:
This study will compare 2 methods to clean contaminated implant surfaces: air-polishing device versus titanium curette. Both of these methods will be used in the non-surgical and surgical setting, followed by implant removal. Then, in-vitro analysis to assess the efficacy of surface decontamination will be performed.

DETAILED DESCRIPTION:
A screening visit will be performed to determine the elegibility of the individuals to participate in the study. Information related to the target implant (e.g., brand, material, surface, dimensions, time of function, history of treatment of peri-implantitis) and reconstruction (e.g., cemented or screwed prosthesis, single, multi-unit or full-arch) will be collected. Intra-oral radiographs will be obtained or exported from patients' dental records, and the marginal bone level (MBL) will be measured at the mesial and distal aspects of the implants by one calibrated investigator using an image analysis software (Image J; National Institutes of Health, Bethesda, MD, USA). The anatomy of the bone defect will be determined.

Randomization will be performed in a stratified manner, in sets of 10 implants, by a computer software, to obtain equally balanced groups based on implant characteristics (site, brand, design). A researcher not involved in the clinical interventions will be responsible for randomization.

At the day of implant removal, a single calibrated examiner will assess the following parameters at six sites around each experimental implant using an UNC 15 periodontal probe: (1) Plaque accumulation, using the modified plaque index [mPI]; (2) Probing depth (mm); (3) Bleeding on probing, using the modified gingival index [mGI] ; (4) Suppuration; (5) Recession (mm). The width of keratinized mucosa (KM) will be obtained in the mid-buccal and mid-lingal aspect of the implants (mm). A standard tessellation language (STL) file of the arch of interest using an intraoral optical scanner (Trios 3, 3Shape, Denmark) will be obtained.

Surface decontamination protocols:

All cleaning procedures will be performed without the suprastructures. A notch will be performed on the buccal side of all implant shoulders with the aid of a bur, in order to distinguish the different implant surfaces during the microbiological and biocompatibility analysis phases.

Following local anesthesia, implants will be randomly assigned to the following study groups:

1. Non-surgical decontamination with titanium curettes prior to implant removal (n = 20);
2. Non-surgical decontamination with erythritol powder prior to implant removal (n = 20);
3. Surgical decontamination with titanium curettes prior to implant removal (n = 20);
4. Surgical decontamination with erythritol powder prior to implant removal (n = 20);
5. No decontamination prior to implant removal (n=10).

In the surgical groups, intra-sulcular and, if necessary, vertical releasing incisions will be performed. Full-thickness flaps will be elevated in the buccal and lingual aspects and the granulation tissue will be removed.

All giant (visible) calculus will be removed with an ultrasonic tip in advance, without touching the implant surface directly. Copious irrigation with saline will be performed in both groups prior to implant decontamination. All implants will be cleaned by the same operator with the aid of dental surgical loupes. The time needed for the operator to consider the implant surface clean will be recorded.

* Titanium curettes (Hu-Friedy, Chicago, Illinois, USA) will be used for supra and submucosal around the implants.
* Air-polishing (Airflow Prophylaxis Master, EMS, Nyon, Switzerland) will be carried out with AIR-FLOW powder PLUS (EMS) containing erythritol (sugar alcohol, 14 μm), amorphous silica and 0.3% chlorhexidine. The device will be adjusted to a power setting of 5 bar static pressure and a maximum level of irrigation with water.

  * Non-surgical group: The supramucosal implant surfaces will be cleaned with the Airflow handpiece, while for the submucosal areas, a Perioflow handpiece and nozzle for submucosal instrumentation will be used. The nozzle will be changed after cleaning each implant.
  * Surgical group: The Airflow handpiece will be moved in a horizontal direction along implant threads from an apical to a coronal position. The angulation of the handpiece and working distance will not be standardized as they may vary according to the area being cleaned.

Implant removal:

Once the decontamination procedure has been completed, all the implants will be explanted with the aid of a reverse torque device (Implant Removal Kit; Zimmer Biomet); no trephines will be used. During the procedure, care will be taken to avoid damage to the implant and its surface. The retrieved implants will be immersed in a transport medium (Dulbecco's Modified Eagle Medium) and stored in sterile plastic vials at 4°C until further analysis.

In all study groups, the explanted sites will be again curetted and the soft tissues will be sutured with interrupted or crossed sutures. Subjects will receive detailed verbal and written postoperative instructions, as well as a prescription for anti-inflammatory medication (ibuprofen [600mg], for 3-5 days, as needed for pain control). Patients will be instructed to rinse gently with 0.12% chlorhexidine twice daily for 1 week. Sutures will be removed after 2 weeks.

Subsequently, a second randomization will take place to direct each implant (n = 10 in each decontamination group) for microbiological/elementary composition analysis and biocompatibility analysis. In-vitro analysis post surface decontamination includes assessing the cleaning efficacy, microbiological analysis, biocompatibility analysis including cultivation of cells, RNA extraction, Reverse Transcription (RT) and Real-Time RT-Polymerase Chain Reaction (Real-Time RT-PCR) , and elementary composition analysis including implant surface degradation, corrosion performance and atomic composition.

ELIGIBILITY:
Inclusion criteria:

* Adult individuals between 18 and 80 years of age who require the explantation of at least one titanium or titanium alloy implant due to severe peri-implantitis (> 50% bone loss and signs of inflammation);
* Individuals who did not undergo surgical or non-surgical peri-implant therapy in the previous 6 months.

Exclusion criteria:

* Acute infection associated with adjacent teeth;
* Any technical complication that does not allow implant removal using a reverse torque device;
* Active infectious diseases of any kind;
* Medical conditions which requires premedication prior to dental treatments/visits;
* Pregnant women or planning to become pregnant (self-reported);
* History of radiotherapy in the head and neck or chemotherapy in the last 3 years;
* Any other diseases or medications that may contraindicate the surgical procedure or compromise wound healing.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-05-21 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of clean implant surface area following implant decontamination approaches | Right after decontamination and implant removal (T0)
  The cleaned surface area will be planimetrically recorded, and the percentage presence/absence of mineralized deposits as well as scratches on the decontaminated implant surfaces will be determined with the aid of a stereomicroscope.

SECONDARY OUTCOMES:
Bacterial composition of the implants | Right after decontamination and implant removal (T0)
  Shotgun metagenomic sequencing will be used to identify the bacterial composition in the residual biofilms.
Biocompatibility analysis of the implant | Right after decontamination and implant removal (T0)
  Cultivation of osteoblastic cells will be performed and assessed on the implants.
Scanning electron microscopy analysis of the cells and residual bacterial deposits | Right after decontamination and implant removal (T0)
  SEM images of the surfaces of negative control implants (brand new) and treated implants for each decontamination method will be exemplarily taken after instrumentation and cell culture.
Patient satisfaction with the decontamination devices | Right after decontamination and implant removal (T0)
  Patients will be asked to fill out a questionnaire.
Incidence of complications | Right after decontamination and implant removal (T0)
  Incidence of complications will be recorded by the clinician performing the intervention.
Implant surface degradation | Right after decontamination and implant removal (T0)
  Three-dimensional images and roughness line profiles will be acquired by laser scanning confocal microscopy.
Corrosion performance | Right after decontamination and implant removal (T0)
  In vitro electrochemical tests will be conducted to determine the corrosion performance.
Atomic composition of the implants after removal | Right after decontamination and implant removal (T0)
  The atomic composition of the surface of the decontaminated implants will be examined using energy-dispersive x-ray spectroscopy (EDS).

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Ravida, DDS MS PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, School of Dental Medicine, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No